CLINICAL TRIAL: NCT01797341
Title: Prograf/Advagraf Conversion Study in Kidney Pancreas Transplant Recipients
Brief Title: Prograf-Advagraf Cross Over Conversion Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-0330-B
Record Dates: First submitted 2013-02-11; First posted 2013-02-22 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-07

CONDITIONS: Kidney-Pancreas Transplantation
Keywords: Renal Transplantation; Kidney transplantation; Pancreas Transplantation; Tacrolimus; Advagraf; Prograf; Drug Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf arm (Experimental): patients will self-administer tacrolimus in the form of Prograf (twice daily administration.
  Dosage will be adjusted to maintain trough serum levels of 5-15 μg/ml. Maximum daily dose of 20 mg once per day.
  Interventions: Drug: Tacrolimus
- Advagraf Arm (Experimental): patients will self-administer tacrolimus in the form of Advagraf (once daily dosing) Dosage will be adjusted to maintain trough serum levels of 5-15 μg/ml. Maximum daily dose of 20 mg once per day.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus
  Other Names: Prograf
  Arms: Prograf arm
Drug: Tacrolimus
  Other Names: Advagraf
  Arms: Advagraf Arm

SUMMARY:
The present study is aimed at evaluating the impact of a switch from Prograf to Advagraf on renal function, trough tacrolimus levels, drug-related adverse effects and adherence in stable recipients of kidney-pancreas transplants. MPA pharmacokinetics will also be evaluated. The results of this study have the potential to change current practice.

DETAILED DESCRIPTION:
Tacrolimus (Prograf ©) has become part of the standard of care for patients receiving solid organ transplants and is part of the immunosuppressive protocol used by kidney-pancreas transplant recipients at University Health Network (UHN). Tacrolimus is associated with several toxicities, and as a result, careful therapeutic drug monitoring of tacrolimus is a key component of post-transplant management. Trough serum concentrations of tacrolimus are measured routinely and are used to guide dosing. Tacrolimus trough levels are known to correlate with total drug exposure. The Prograf formulation of tacrolimus has a fairly short serum half-life and must be dosed twice daily to maintain therapeutic serum concentrations. This results in two high peak levels each day which have been shown to correlate with toxicity. Thus, avoidance of high peaks may be desirable to minimize tacrolimus toxicity.

Advagraf is a new preparation of tacrolimus that is formulated to provide similar drug exposure to tacrolimus but with a once daily dosing regimen, which avoids the 2 daily high tacrolimus peaks observed with Prograf. In this way, it is hoped that Advagraf may provide similar therapeutic efficacy as Prograf but with fewer adverse effects. In addition, the simpler dosing regimen is expected to enhance patient adherence. Tacrolimus has also been shown, along with many other drugs, to have a variable impact on mycophenolate acid (MPA) pharmacokinetics. There are currently few data on whether Advagraf impacts MPA pharmacokinetics to the same or a lesser degree than Prograf.

Eligible kidney-pancreas recipients will be recruited and after obtaining informed consent, randomized to continue their current total daily Prograf dosage or switch to the equivalent once daily dose of Advagraf. Patients will continue randomized therapy for 12 weeks and will then cross over to the opposite therapy for another 12 weeks. Patients will be followed and maintained on the same medication designated at week 24. Bloodwork results, adherence and AEs (adverse events) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* recipient of kidney and pancreas transplant
* aged 18 years or older
* 12 months or more since time of transplant
* stable allograft function (creatinine < 180 µmol/l and eGFR > 40 ml/min)
* targeted to a tacrolimus trough level of 5-10 ug/ml that has been stable during the prior 3 mo.

Exclusion Criteria:

* episode of acute rejection within 6 months of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Tacrolimus trough levels | prior to conversion and 12 weeks post-conversion
  Serum trough levels
Change in Renal Function | prior to conversion and 12 weeks post-conversion
  Serum creatinine and urea levels
Change in Tacrolimus dosage (week 12 compared to week 24) | week 12 and week 24

SECONDARY OUTCOMES:
Change in Fasting glucose | prior to conversion and 12 weeks post-conversion
  serum fasting glucose levels
Lipid profile | prior to conversion and 12 weeks post-conversion
  Cholesterol, etc...
blood pressure | prior to conversion and 12 weeks post-conversion
  Cuff blood pressure readings
Drug Adherence | assessed at weeks 12 and 24
  patient self-reported drug adherence
Number of Participants with Adverse Events as a Measure of Safety and Tolerability" | at week 12 and week 24
  at every visit, patients will be asked about and assessed for any adverse event development

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Cattral, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada